CLINICAL TRIAL: NCT01324076
Title: TACE-2: A Randomized Placebo-Controlled, Double Blinded, Phase III Trial of Sorafenib in Combination With Transarterial Chemoembolization in Hepatocellular Cancer
Brief Title: Transarterial Chemoembolization Using Doxorubicin Beads With or Without Sorafenib Tosylate in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000697324; CRUK-TACE-2; UCL-07130; EU-21108; CRUK-HE3005; EUDRACT-2008-005073-36; CRUK-13136; ISRCTN-93375053; CTA-20363/0272/001; BAYER-CRUK-TACE-2; BIOCOM-UK-CRUK-TACE-2
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib; Pharmacogenomic Testing

INTERVENTIONS:
Drug: doxorubicin-eluting beads
Drug: sorafenib tosylate
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Other: pharmacological study
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by carrying drugs directly into the tumor and blocking the blood flow to the tumor. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether transarterial chemoembolization using doxorubicin-eluting beads is more effective when given with or without sorafenib tosylate in treating patients with liver cancer that cannot be removed by surgery.

PURPOSE: This randomized phase III trial is studying giving transarterial chemoembolization using doxorubicin-eluting beads and sorafenib tosylate to see how well it works compared with giving transarterial chemoembolization using doxorubicin-eluting beads and a placebo in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the addition of sorafenib tosylate to transarterial chemoembolization (TACE) with doxorubicin-eluting beads, compared to TACE alone, prolongs progression-free survival of patients with unresectable hepatocellular carcinoma.

Secondary

* To determine if adding sorafenib tosylate to TACE prolongs overall survival of these patients.
* To determine if the sorafenib tosylate regimen prolongs time to progression in these patients.
* To determine acceptable toxicity related to the sorafenib tosylate regimen in these patients.
* To determine the effects of the sorafenib tosylate regimen on disease response, in terms of complete response, partial response, or stable disease, in these patients.
* To determine the effects of the sorafenib tosylate regimen on quality of life of these patients.
* To determine if treatment with the sorafenib tosylate regimen reduces the frequency for repeat TACE as measured by number of TACE procedures performed in 12 months.
* To establish a blood sample bank linked to this study for biomarker research (proteomic and genomic analysis).

OUTLINE: This is a multicenter study. Patients are stratified according to randomizing centers and serum alpha-fetoprotein levels (< 400 ng/mL vs ≥ 400 ng/mL). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate twice daily in the absence of disease progression or unacceptable toxicity. Beginning within 2-5 weeks after start of sorafenib tosylate, patients undergo transarterial chemoembolization (TACE) with doxorubicin-eluting beads. Patients may undergo additional sessions of TACE with doxorubicin-eluting beads, in the absence of complete devascularization of the tumor(s) (as assessed by follow-up contrast enhanced scan).
* Arm II: Patients receive oral placebo twice daily in the absence of disease progression or unacceptable toxicity. Beginning within 2-5 weeks after start of placebo, patients undergo TACE with doxorubicin-eluting beads as in arm I. Patients with disease progression may cross over to the sorafenib tosylate arm at the discretion of the treating clinician and are followed for survival.

Blood samples may be collected at baseline and periodically for pharmacogenetic and pharmacokinetic studies. Patients complete EORTC QoL questionnaire (QLQ-C30) version 3 and EORTC QLQ-HCC18 (a site-specific module for HCC) at baseline and periodically during the study.

After completion of study therapy, patients are followed up periodically for 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC) OR meets the American Association for the Study of Liver Diseases (AASLD) criteria for diagnosis of HCC

  * Unresectable disease
  * Not amenable to liver transplantation
* At least one uni-dimensionally measurable lesion according to the RECIST criteria by CT scan or MRI
* Child-Pugh A (score ≤ 6) and no Child-Pugh cirrhosis C or B (score ≥ 7)
* No ascites refractory to diuretic therapy
* No documented occlusion of the hepatic artery or main portal vein
* No extrahepatic metastasis or hepatic encephalopathy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* Hemoglobin ≥ 9 g/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 60,000/μL
* Bilirubin ≤ 50 μmol/L
* Alkaline phosphatase < 4 times upper limit of normal (ULN)
* AST and ALT < 5 times ULN
* Creatinine ≤ 1.5 times ULN
* Amylase and lipase < 2 times ULN
* INR ≤ 1.5
* LVEF ≥ 45%
* Able to swallow oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for 3 months after completion of study treatment
* No history of bleeding within the past 4 weeks
* No contraindications for hepatic embolization procedures, including portosystemic shunt, hepatofugal blood flow, or known severe atheromatosis
* No hypersensitivity to intravenous contrast agents
* No active clinically serious infection > grade 2 (NCI-CTC version 4)
* No known history of HIV infection
* No history of second malignancy except non-melanotic skin cancer or cervical carcinoma in situ or malignancy treated with curative intent with > 3 years without relapse
* No evidence of severe or uncontrolled disease including any of the following:

  * Systemic disease
  * Cardiac arrhythmias (requiring anti-arrhythmic therapy or pacemaker)
  * Hypertension
  * NYHA class III or IV congestive cardiac failure
  * Myocardial infarction within the past 6 months
  * Laboratory finding that, in the view of the Investigator, makes it undesirable for the patient to participate in the trial
* No psychiatric or other disorder likely to impact on informed consent

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior and no concurrent investigational therapy
* No prior embolization, systemic therapy, or radiotherapy for HCC
* No major surgery within the past 4 weeks
* No ablative therapy (radiofrequency ablation or percutaneous ethanol injection) for HCC

  * Patients with untreated target lesion(s) and ablation occurred > 6 weeks prior to study entry allowed
* No concurrent rifampicin or St. John wort
* No concurrent bone marrow transplant or stem cell rescue
* No concurrent bevacizumab or drugs that target VEGF or VEGF receptors
* No other concurrent anticancer chemotherapy, immunotherapy, hormone therapy, or molecular therapy except bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Time to progression
Toxicity
Disease control (complete or partial response or stable disease)
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, MD, BSc, MRCP, PhD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Bristol Royal Infirmary, Bristol, England
  - Aintree University Hospital, Liverpool, England
  - Royal Free Hospital, London, England
  - King's College Hospital, London, England
  - Royal Marsden - London, London, England
  - Queen's Medical Centre, Nottingham, England
  - Southampton General Hospital, Southampton, England